CLINICAL TRIAL: NCT03085641
Title: Treatment of Central Sleep Apnoea and Cheyne Stokes Respiration in Patients With Heart Failure: Nasal High-flow Oxygen Therapy?
Brief Title: Treatment of Central Sleep Apnoea in Patients With Heart Failure With Nasal High Flow Therapy (nHFT)
Acronym: RELAX
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Side effects
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Marieke Duiverman, Pneumologist, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201700147
Record Dates: First submitted 2017-03-08; First posted 2017-03-21 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Central Sleep Apnea; Cheyne-Stokes Respiration
Keywords: High flow oxygen therapy
MeSH Terms: conditions — Sleep Apnea, Central; Cheyne-Stokes Respiration

STUDY DESIGN:
Intervention Model Description: prospective one armed uncontrolled intervention pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nasal high flow oxygen therapy (Experimental): The patient is hospitalized for one night.
  Initially patients will start with a flow rate of 10 L/min and when they are asleep during the night 90-minute periods of the following settings will be performed:
  * Moderate flow rate: 20 L/min without additional oxygen (with room air, which means a fractional inspired oxygen (FiO2) of 21%)
  * High flow rate: 40-50 L/min without additional oxygen
  * Moderate flow rate: 20 L/min with FiO2 of 28% (comparable to the 2 L/min additional oxygen through a nasal cannula)
  * High flow rate: 40-50 L/min with FiO2 of 28%
  Interventions: Device: Nasal high flow oxygen therapy

INTERVENTIONS:
Device: Nasal high flow oxygen therapy — nHFT will be titrated during a first titration night and used at home during the night for 4 weeks consecutively

SUMMARY:
To investigate whether nHFT is an effective treatment for patients with Chronic Heart Failure (CHF) and central sleep apnea (CSA).

This study is a prospective one armed uncontrolled intervention pilot study investigating 4 weeks of nHFT at home in 10 patients with CHF and CSA.

DETAILED DESCRIPTION:
Study population: 10 CHF patients with a Left Ventricular Injection Fraction(LVEF)< 45% and CSA/Cheyne Stokes Respiration (CSR) (apnoea/hypopnea index (AHI) > 15/hour); with at least 50% of the total number of events having a central character will be included. Patients with other diseases that will influence the respiratory system negatively during sleep i.e. chronic obstructive pulmonary disease (COPD Global Initiative of Obstructive Lung Diseases (GOLD) class 3 and 4), neuromuscular diseases and thorax cage deformities, as well as patients with CHF and CSA that use another form of treatment for their CSA at the time of inclusion, will be excluded.

Intervention: nHFT will be titrated during a first titration night and used at home during the night for 4 weeks consecutively.

Main study parameters/endpoints:

1. To investigate the effect of nHFT with and without oxygen in reducing the apnoea/hypopnoea index during sleep after 4 weeks use nHFT.
2. To investigate improvements in oxygen desaturation index, sleep quality and sleepiness, physical condition, left ventricular ejection fraction (LVEF), heart beat variability (HRV), N-terminal natriuretic peptide (NTproBNP) after 4 weeks use nHFT .
3. Physiological condition; work of breathing and respiratory drive and measuring mouth-throat pressure.

ELIGIBILITY:
Inclusion Criteria:

1. Moderate to severe CSA/CSR (AHI>15), in which CSA is defined when at least 50% of the apnoeas are central apnoeas
2. Heart failure with reduced ejection fraction, defined as a LVEF < 45% of predicted

Exclusion Criteria:

1. Other diseases affecting respiration during sleep (COPD GOLD 3 or 4, neuromuscular disorders, thorax cage deformities)
2. At the moment of the inclusion, the patient does not have a therapy to treat the CSA, such as continuous positive airway pressure (CPAP), oxygen, bilevel intermittent positive airway pressure (BiPAP) or acetazolamide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2018-10-18 (Actual)

PRIMARY OUTCOMES:
Reduction of apnea/hypopnea index | Baseline, 4 weeks
  the change/reduction in AHI after 4 weeks of treatment with nHFT.

SECONDARY OUTCOMES:
Improvement physical condition | Baseline, 4 weeks
  Exercise tolerance assessed with the 6-minute walking test
Work of breathing | Baseline titration night
  Transdiaphragmatic pressure as a marker of diaphragmatic true work of breathing, measured with the use of oesophageal and gastric balloon catheters
Drive to breath | Baseline titration night, 4 weeks
  Drive to breath assessed with surface electromyography (EMG) of the respiratory muscles
Sleep latency | Baseline, 4 weeks
  Assessed as the the length of time that it takes to accomplish the transition from full wakefulness to sleep, measured by means of electro-encephalogram (ECG) as part of the polysomnography
Cardiac functioning | Baseline, 4 weeks
  Left ventricular injection fraction (LVEF),
change in oxygen desaturation index (ODI) during sleep while on nHFT | Baseline, 4 weeks
  measured after 4 weeks of home nHFT treatment, as compared to the baseline ODI during spontaneous nocturnal breathing.
Sleep efficiency | Baseline, 4 weeks
  The percentage of total time in bed actually spent in sleep, assessed with polysomnography
Total rapid-eye movement (REM) stage sleep cycles recorded | Baseline, 4 weeks
  Assessed with polysomnography
Heart rate variability | Baseline, 4 weeks
  Heart rate variability will be assessed by 24-uur ECG recordings
N-terminal natriuretic peptide (NTproBNP) | Baseline, 4 weeks
  Assessed in venous blood

CONTACTS AND LOCATIONS:
Overall Officials: Marieke Duiverman, Study Director — University Medical Center Groningen
Locations (1):
- Department of Pulmonary diseases, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No